CLINICAL TRIAL: NCT01216319
Title: A Single Arm Multicenter Study Evaluating the Cook Biodesign® Nipple Reconstruction Cylinder (NRC)
Brief Title: Evaluation of the Cook Biodesign® Nipple Reconstruction Cylinder (NRC)
Acronym: NRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-009
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Breast Reconstruction; Nipple Reconstruction
Keywords: Biodesign; Nipple Reconstruction; Breast Cancer; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Nipple Reconstruction Cylinder (Experimental)
  Interventions: Device: Nipple reconstruction

INTERVENTIONS:
Device: Nipple reconstruction — Biodesign® Nipple Reconstruction Cylinder
  Other Names: Biodesign

SUMMARY:
Patients with a desire for nipple reconstruction following breast cancer and breast reconstruction will receive a surgical procedure to reconstruct one or both nipples utilizing the COOK Biodesign® Nipple Reconstruction Cylinder.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with a history of breast cancer, having previously completed either uni- or bi-lateral breast removal and reconstruction.
* Patient presents with a desire to obtain nipple reconstruction
* Patient is at least 18 years of age
* And other inclusion criteria

Exclusion Criteria:

* Patient is not medically fit enough for surgery under local anesthesia
* Patient is currently smoking, using tobacco products, or nicotine products (i.e. patch, gum, or nasal spray)
* Patient is pregnant, breastfeeding or planning further pregnancy during the study period
* Patient has physical allergies or cultural objections to the receipt of porcine products
* And other exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Gurtner, MD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Park Meadows Cosmetic Surgery, Lone Tree, Colorado
  - Mercy Medical Center, Baltimore, Maryland
  - Sanford Clinic Plastic and Reconstructive Surgery, Sioux Falls, South Dakota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nipple Reconstruction Cylinder
Started | 50
Completed | 46
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Unanticipated chemo for breast cancer | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nipple Reconstruction Cylinder
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Nipple Projection at 12 Months Compared to Baseline (1 Week Post-procedure)
Time Frame: 12 months
Population: There were two patients (three nipples) without plastic surgery matrix in place at 12MO.
Measure: Mean (Standard Deviation); unit: percentage of projection vs baseline
Units Other Than Participants: Nipples
Arm/Group | Nipple Reconstruction Cylinder
Number analyzed (Participants) | 44
Number analyzed (Nipples) | 72
percentage of projection vs baseline | 37.3 (17.5)

2. Secondary Outcome: Rate of Patient Satisfaction
Description: Patient satisfaction is defined as patient would recommend the nipple reconstruction operation to others.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Nipple Reconstruction Cylinder
Number analyzed (Participants) | 46
percentage of patients | 97.8

ADVERSE EVENTS:
Arm/Group | Nipple Reconstruction Cylinder
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nipple Reconstruction Cylinder (N=50)
Metastatic breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nipple Reconstruction Cylinder (N=50)
Cylinder extrusion (Surgical and medical procedures) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days